CLINICAL TRIAL: NCT04975334
Title: Opioid Antagonism in Hypogonadotropic Hypogonadism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stephanie B. Seminara, MD (Other)
Responsible Party: Sponsor-Investigator, Stephanie B. Seminara, MD, Chief, Reproductive Endocrine Unit; Professor of Medicine, Harvard Medical School; Director, MGH Harvard Center for Reproductive Medicine, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 313510
Record Dates: First submitted 2021-07-15; First posted 2021-07-23 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Hypogonadotropic Hypogonadism; Low Testosterone
Keywords: Hypogonadotropic Hypogonadism; naloxone
MeSH Terms: conditions — Hypogonadism | interventions — Naloxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- naloxone (Experimental): one period of frequent blood sampling with IV administration of naloxone (one bolus)
  Interventions: Drug: Naloxone

INTERVENTIONS:
Drug: Naloxone — One bolus of naloxone

SUMMARY:
The goal of this study is to evaluate the effects of opioid antagonists on the hypothalamic-pituitary-gonadal axis in subjects with hypogonadotropic hypogonadism (HH).

DETAILED DESCRIPTION:
Assignment: Each study subject will serve as their own control.

Delivery of Interventions:

* Prior to the study visit, subjects will undergo a review of their medical history and screening laboratories.
* During the study, the subjects will undergo the following:

  * Undergo q10 min blood sampling for 3 hours
  * Receive a naloxone bolus at the midpoint of q10 min sampling

ELIGIBILITY:
Inclusion

* Male
* Age 18-75 years
* Confirmed diagnosis of hypogonadotropic hypogonadism (low testosterone)
* All medical conditions stable
* Normal blood pressure (systolic BP < 140 mm Hg, diastolic < 90 mm Hg)
* Negative urine drug screening panel
* Hemoglobin
* Men on adequate testosterone replacement therapy: normal male reference range
* Men off testosterone replacement therapy: no lower than 0.5 gm/dL below the lower limit of the reference range for normal women

Exclusion

* Any condition (medical, mental, or behavioral) that, in the opinion of a study investigator, would likely interfere with participation in/completion of the protocol
* Current or recent use of a medication (including hormonal replacement) that, in the opinion of a study investigator, can modulate the reproductive axis and, if applicable, unwilling to complete an appropriate washout for that particular medication and its method of administration
* Current or recent use of a medication that affects the opioid pathway
* Active illicit drug use

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2025-06-18 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Average change in mean Luteinizing Hormone (LH) value | Before and after treatment
  Change in mean LH before vs. after naloxone bolus

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Seminara, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No